CLINICAL TRIAL: NCT01615289
Title: Neural Effects of Green Tea Extract on Dorsolateral Prefrontal Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christoph Beglinger, Professor of Medicine, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EKBB 32/09
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Exploratory Behavior
MeSH Terms: conditions — Exploratory Behavior | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Green tea extract, 250 ml (Active Comparator): Single intragastric instillation of 250 ml green tea extract
  Interventions: Dietary Supplement: Single intragastric instillation of 250 ml green tea extract
- Green tea extract, 500 ml (Active Comparator): Intragastric instillation of 500 ml green tea extract solution
  Interventions: Dietary Supplement: Single intragastric instillation of 500 ml green tea extract
- Control solution, 250 ml (Placebo Comparator): Intragastric instillation of 250 ml control solution
  Interventions: Dietary Supplement: Single intragastric instillation of 250 ml control solution
- Control solution, 500 ml (Placebo Comparator): Single intragastric instillation of 500 ml control solution
  Interventions: Dietary Supplement: Single intragastric instillation of 500 ml control solution

INTERVENTIONS:
Dietary Supplement: Single intragastric instillation of 250 ml green tea extract — Intragastric instillation by feeding tube
  Arms: Green tea extract, 250 ml
Dietary Supplement: Single intragastric instillation of 500 ml green tea extract — Intragastric instillation by feeding tube
  Arms: Green tea extract, 500 ml
Dietary Supplement: Single intragastric instillation of 250 ml control solution — Intragastric instillation by feeding tube
  Arms: Control solution, 250 ml
Dietary Supplement: Single intragastric instillation of 500 ml control solution — Intragastric instillation by feeding tube
  Arms: Control solution, 500 ml

SUMMARY:
Green tea is being recognized as a beverage with potential benefits for human health and on cognitive function. In vitro and in vivo studies provide preliminary evidence that green tea intake may play a positive role in improving effects on cognitive functions. The investigators aim to examine the neural effects of green tea extract on brain activation in humans.

DETAILED DESCRIPTION:
As functional neuroimaging provides a means of examining how green tea extract acts on the brain, we used functional magnetic resonance imaging (fMRI) to study healthy volunteers while they performed a working memory task following intra-gastric administration of either 250 ml or 500 ml Rivella green® (RG), a milk whey based green tea extract containing soft drink, or Rivella blue® (RB), a milk whey based soft drink without green tea extract as sham condition in a double-blind, controlled design. Based on the literature on pharmacological and behavioural effects of green tea, we hypothesized - a priori - that green tea extract would subtly modulate the engagement of the dorsolateral prefrontal cortex (DLPFC), a brain region critically involved in many cognitive functions such as working memory processing.

A double-blind, controlled, within-subject study with counterbalanced order of substance administration using an established protocol (6-8) was conducted over 4 sessions (250 ml or 500 ml Rivella green® (including green tea extract; RG), 250 or 500 ml Rivella blue® (RB). Each participant was scanned four times with a one-week interval between scans. The order of substance administration across sessions was counterbalanced across subjects, such that equal numbers followed each substance sequence.

ELIGIBILITY:
Inclusion Criteria:

* right-handed healthy males, no drugs, non-smoking

Exclusion Criteria:

* drug abuse, smoker, left-handed

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) in healthy volunteers while they performed a working memory task | 0 and 45 min
  Whole brain analysis with a cluster-level threshold was followed by an a priori defined region of interest analysis of the dorsolateral prefrontal cortex including a cluster-level threshold and family-wise error adjustment for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland